CLINICAL TRIAL: NCT01041612
Title: Prospective Randomized Trial Comparing Covered Metal Stents Placed Above and Across the Sphincter of Oddi in Malignant Biliary Obstruction: A Multi-nation, Multi-center Study
Brief Title: Comparing Covered Self-expandable Metallic Stent (SEMS) Above/Across the Sphincter of Oddi
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Taewoong Medical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Jong Taek, Lee, General manager, Taewoong Medical Co., Ltd.
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: RaMM-BO 2.0
Record Dates: First submitted 2009-12-28; First posted 2010-01-01 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-10

CONDITIONS: Cancer of Bile Duct; Pancreatic Cancer
Keywords: CBD; HBD; cancer of bile duct; pancreatic cancer
MeSH Terms: conditions — Bile Duct Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A: C-SEMS, inserted above SO (Active Comparator): -In group A, SO should be preserved without sphincterotomy, but small infundibulotomy with needle knife can be accepted for cannulation.
  Interventions: Device: PTFE Covered ComVi [full covered] Biliary Stent
- Group B: C-SEMS, inserted across SO (Active Comparator): -In group B, small sphincterotomy (50% incision) will be done after biliary cannulation.
  Interventions: Device: PTFE Covered ComVi [full covered] Biliary Stent

INTERVENTIONS:
Device: PTFE Covered ComVi [full covered] Biliary Stent — The stent is made of Nitinol wire. It is a flexible, fine mesh tubular prosthesis and it has 10 radiopaque markers; 4 in each end and 2 in the center.
  Other Names: PTFE Covered ComVi [full covered] Biliary Stent, Taewoong Medical, Korea
  Arms: Group A: C-SEMS, inserted above SO
Device: PTFE Covered ComVi [full covered] Biliary Stent — The stent is made of Nitinol wire. It is a flexible, fine mesh tubular prosthesis and it has 10 radiopaque markers; 4 in each end and 2 in the center.
  Other Names: PTFE Covered ComVi [full covered] Biliary Stent, Taewoong Medical, Korea
  Arms: Group B: C-SEMS, inserted across SO

SUMMARY:
The purpose of this prospective, randomized multicenter study is to determine whether there is any difference in stent patency of covered metallic stents in terms of stent positioning, above and across the sphincter of Oddi, in malignant bile duct obstruction.

ELIGIBILITY:
Inclusion Criteria:

* Inoperable and/or unresectable cases of malignant stenosis at distal common hepatic duct or CBD, >= 18 years old
* Bile duct or gallbladder cancer invading CBD or distal CHD
* Pancreatic cancer with mid or distal CBD invasion
* Cancer should be 1.5 cm apart from bifurcation and 2 cm apart from ampulla of Vater.
* First attempt of endoscopic biliary metallic stenting
* Negative history of biliary tract surgery
* Life expectancy at least longer than 4 months (Karnofsky score >60%)

Exclusion Criteria:

* Ampullary cancer
* Klatskin tumor
* Combined intrahepatic bile duct cancer
* Patient with hemobilia
* Previous history of biliary drainage (endoscopic, percutaneous, surgical) except plastic stent or endoscopic nasobiliary drainage smaller than 7 Fr within 14 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-01; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Obstruction of 1st C-SEMS or presence of jaundice at death without stent exchange | one year

SECONDARY OUTCOMES:
Death of patients | one year

CONTACTS AND LOCATIONS:
Overall Officials: Dong Ki Lee, PH.D, Principal Investigator — Gangnam Severance Hospital
Locations (13):
- Japan (7):
  - Gifu University, Gifu
  - Onomichi General Hospital, Onomichi
  - Teine-Keijinkai Hospital, Sapporo
  - The University of Tokyo, Tokyo
  - Toho University, Tokyo
  - Tokyo Medical University, Tokyo
  - Yamaguchi University, Ube
- South Korea (6):
  - Soon Chun Hyang University School of Medicine, Bucheon-si
  - Soon Chun Hyang University School of Medicine, Cheonan
  - Catholic University of Daegu School of Medicine, Daegu
  - Inha University School of Medicine, Incheon
  - Gangnam Severance Hospital, Seoul
  - Ajou University School of Medicine, Suwon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jung Nam Cho, Jimin Han, Ho Gak Kim, IM Hee Shin, Sang Heum Park, Jong Ho Moon, Jin Hong Kim, Don Haeng Lee, Iruru Maetani, Hiroyuki Maguchi, Keiji Hanada, Ichiro Yasuda, Takao Itoi, Hiroyuki Isayama, Dongki Lee. Prospective Randomized Trial Comparing Covered Metal Stent Placed Above and Across the Sphincter of Oddi in Malignant Biliary Obstruction. Gastrointestinal Endoscopy 77(58): AB139-AB140, 2013